CLINICAL TRIAL: NCT00389090
Title: A Phase II Study of Temozolomide and O6-Benzylguanine (O6-BG) in Patients With Temozolomide-Resistant Anaplastic Glioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: AOI Pharma terminated the license agreement. IND Transferred to NCI
Sponsor: Keryx / AOI Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: O6BG 202
Record Dates: First submitted 2006-10-16; First posted 2006-10-18 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Glioma; Astrocytoma; Oligodendroglioma; Oligoastrocytoma
Keywords: temozolomide resistant; anaplastic glioma; anaplastic astrocytoma; anaplastic oligodendroglioma; anaplastic oligoastrocytoma
MeSH Terms: conditions — Glioma; Astrocytoma; Oligodendroglioma | interventions — Temozolomide; O(6)-benzylguanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temozolomide + O6BG (Experimental)
  Interventions: Drug: Temozolomide and O6-Benzylguanine

INTERVENTIONS:
Drug: Temozolomide and O6-Benzylguanine — O6BG + Temozolomide
  Other Names: temodar

SUMMARY:
This is an open-label, multicenter, phase II trial, assessing the antitumor activity, and safety of temozolomide in combination with O6-BG in patients with temozolomide-resistant anaplastic glioma.

DETAILED DESCRIPTION:
This open-label, multicenter, phase II trial will assess the antitumor activity and safety of temozolomide in combination with O6-BG in patients with temozolomide-resistant anaplastic glioma.

Forty-one to 104 evaluable patients with temozolomide-resistant anaplastic glioma will be enrolled in this study. Total accrual on this study will not exceed 116 patients. The patients will receive daily temozolomide on 5 consecutive days (days 1-5) along with bolus infusions of O6-BG on days 1, 3, and 5 and a continuous infusion of O6-BG beginning immediately after the first bolus infusion and continuing until immediately prior to the last bolus injection. Patients will be evaluated for AEs during the course of therapy. Patients may receive treatment at the same dose level until appearance of significant treatment-related toxicities, disease progression or withdrawal of consent.

Tumor response will be evaluated at the end of cycle 1, cycle 2 and then every two cycles for the duration of therapy, using physical and neurological examinations and diagnostic imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically documented anaplastic glioma (anaplastic astrocytoma, anaplastic oligodendroglioma or mixed anaplastic oligoastrocytoma).
2. Temozolomide-resistant defined as patients who have progressed while receiving or within 8 weeks of completing the last dose of temozolomide.
3. Disease progression >= 12 weeks after the completion of any radiotherapy.
4. If patient received chemotherapy or an investigational agent as part of their prior therapy, the patient must recover from all toxicities (<= Grade 1) prior to enrollment on this protocol.
5. Bi-dimensionally measurable disease on contrast-enhanced magnetic resonance imaging study (MRI) performed within two weeks of study drug administration.
6. If patient received intratumoral chemotherapy or immunotherapy as part of their prior therapy then histological confirmation of recurrence is mandated.
7. KPS >= 70%.
8. The following laboratory results:

   * Absolute neutrophil count >= 1500 cells/microliter
   * Platelet count >= 100,000 cells/microliter
   * SGOT <= 2.5 x ULN
   * Serum creatinine <= 1.5 x ULN
9. Signed informed consent approved by Institutional Review Board.
10. If sexually active, patients will take contraceptive measures for the duration of the treatment.
11. For patients on corticosteroids, they must have been on a stable dose 1 week prior to baseline MRI and the dose should not be escalated over entry dose level, if clinically possible.

Exclusion Criteria:

1. Pregnant or breast feeding women.
2. Prior treatment with O6-BG plus temozolomide in combination.
3. Active infection requiring intravenous antibiotics.
4. Known diagnosis of Human Immunodeficiency Virus (HIV) infection (HIV testing is not mandatory).
5. Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention.
6. Patients unwilling or unable to comply with the protocol.
7. Patients who have received stereotactic radiosurgery or brachytherapy as part of their prior therapy.
8. Comedication that may interfere with study results; eg. immunosuppressive agents other than corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-10; Primary Completion 2008-06 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
best objective response rate | Month 1, 2 and every 2 months thereafter.

SECONDARY OUTCOMES:
Safety Assessment | Month 1, 2 and every 2 months thereafter
progression-free survival | every 6 months
overall survival | every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Quinn, MD, Study Chair — Preston Robert Tisch Brain Tumor Center at Duke
Locations (12):
- United States (12):
  - AOI Pharmaceuticals Investigative Site, Los Angeles, California
  - AOI Pharmaceuticals Investigative Site, Orlando, Florida
  - AOI Pharmaceuticals Investigative Site, Chicago, Illinois
  - AOI Pharmaceuticals Investigative Site, Evanston, Illinois
  - AOI Pharmaceuticals Investigative Site, Lexington, Kentucky
  - AOI Pharmaceuticals Investigative Site, Louisville, Kentucky
  - AOI Pharmaceuticals Investigative Site, Minneapolis, Minnesota
  - AOI Pharmaceuticals Investigative Site, Durham, North Carolina
  - AOI Pharmaceuticals Investigative Site, Greenville, South Carolina
  - AOI Pharmaceuticals Investigative Site, Dallas, Texas
  - AOI Pharmaceuticals Investigative Site, Houston, Texas
  - AOI Pharmaceuticals Investigative Site, Salt Lake City, Utah